CLINICAL TRIAL: NCT04366011
Title: Efficacy and Mechanisms of Psychosocial Treatments for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Heather McClary, Director of Research Compliance, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011AM/AJ002
Record Dates: First submitted 2013-05-13; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): Cognitive Behavioral Therapy is a twelve-week therapeutic intervention based on the theory that maladaptive thoughts contribute to symptom development and maintenance of PD/A.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Capnometry Assisted Respiratory Training (CART) (Experimental): Capnometry-assisted respiratory therapy is a five-week treatment based on the theory that hyperventilation causes or maintains panic disorder.
  Interventions: Behavioral: Capnometry Assisted Respiratory Training (CART)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT teaches a set of cognitive and somatic coping skills to manage panic and anxiety as patients conduct repeated exposure to feared situations and sensations.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Capnometry Assisted Respiratory Training (CART) — CART has four major treatment components: educating patients about the etiology and maintenance of PD according to a hyperventilation centered rationale, directing patients' attention to potentially aberrant respiratory patterns, instructing patients in respiratory control techniques, and instructing patients in home breathing exercises.
  Arms: Capnometry Assisted Respiratory Training (CART)

SUMMARY:
The aim of the present study is to a) determine the comparative efficacy of the brief capnometry-assisted respiratory therapy (CART) and standard cognitive behavioural therapy (CBT), and b) to determine moderators and mediators.

With the data collected from the study, the investigators will test the following hypotheses: (a) CART will be as effective in treating PD/A as CBT, albeit in shorter time, b) patients with greater respiratory dysregulations, especially hyperventilation, at pretreatment will benefit more from CART, whereas patients with greater cognitive dysregulation will benefit more from CBT. CART, but not CBT, will result in reversal of hyperventilation.

ELIGIBILITY:
Inclusion Criteria:

1. A current DSM-IV (Diagnostic and Statistical Manual IV) diagnosis of panic disorder with or without agoraphobia that is designated by the patient as the most important source of current distress
2. Patients must be willing to engage in exposure to fearful situations and sensations.

Exclusion Criteria:

Diagnostic Exclusion Criteria:

1) A history of bipolar disorder, psychosis or delusional disorders (as evaluated by the SCID-IV-L (Structured Clinical Interview for the DSM IV) screening questions), substance abuse or dependence or alcohol abuse or dependence (other than nicotine in the last 3 months)

Medical exclusion factors:

1. Patients with severe unstable medical illness, clinically significant laboratory findings, or serious medical illness for which hospitalization may be likely within the next three months
2. Patients with a history of seizures, angina, myocardial infarction, congestive heart failure, clinically significant arrhythmias, transient ischemic attacks, cerebrovascular accidents, diabetes mellitus, significant asthma, emphysema, or chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Panic Disorder Symptoms Severity change | During treatment (weeks 1- 12) and 2-months and 6-months follow-ups
  Panic Disorder Severity Scale (PDSS)

SECONDARY OUTCOMES:
End-tidal PCO2 (carbon dioxide partial pressure) change | during treatment (weeks 1-12), 2 -and 6 months follow-up
  End-tidal PCO2

CONTACTS AND LOCATIONS:
Overall Officials: Alicia E Meuret, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- Stress, Anxiety, and Chronic Disease Research Program, Southern Methodist University, Dallas, Texas, United States